CLINICAL TRIAL: NCT02154425
Title: A Multicenter, Postmarketing Study to Evaluate the Concentration of Certolizumab Pegol in the Breast Milk of Mothers Receiving Treatment With Cimzia® (Certolizumab Pegol)
Brief Title: A Multicenter, Postmarketing Study Evaluating the Concentration of Cimzia® in Mature Breast Milk of Lactating Mothers
Acronym: CRADLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP0016; 2013-004126-28 (EudraCT Number)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Axial Spondyloarthritis (AxSpA); Non-radiographic Evidence-AxSpA; Ankylosing Spondylitis; Crohn's Disease; Psoriatic Arthritis; Rheumatoid Arthritis
Keywords: Cimzia®; CZP; Breastfeeding; Nursing; Autoimmune diseases and pregnancy
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Crohn Disease; Arthritis, Psoriatic; Arthritis, Rheumatoid; Breast Feeding; Autoimmune Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetic samples (Experimental): Pharmacokinetic (PK) samples will be taken from breast milk of lactating mothers on an established dosing regimen of CZP on Day 0 of the Sampling Period, just prior to next scheduled dose of CZP, and on Days 2, 4, 6, 8, 10, 12, and 14 (pre-dose if Q2W dosing), relative to CZP administration on Day 0. In addition, in mothers on a CZP Q4W dosing regimen, the concentration of CZP in breast milk will also be evaluated on or about Day 28 (i.e., prior to and on the same day of the next scheduled administration of CZP).
  Included are mothers who decided to continue on, or to start treatment with, Certolizumab Pegol (CZP) for an approved indication with their treating physician prior to participation into this study. The mother is responsible for procuring her own supply of commercial CZP. The CZP dose and administration schedule will be as per the locally approved label.
  Interventions: Procedure: Breast milk sampling; Biological: Certolizumab Pegol

INTERVENTIONS:
Procedure: Breast milk sampling — Pharmacokinetic (PK) samples will be taken from breast milk of lactating mothers on an established dosing regimen of CZP on Day 0 of the Sampling Period, just prior to next scheduled dose of CZP, and on Days 2, 4, 6, 8, 10, 12, and 14 (pre-dose for mothers on CZP Q2W), relative to CZP administration on Day 0. In addition, in mothers on a CZP Q4W dosing regimen, the concentration of CZP in breast milk will also be evaluated on or about Day 28 (i.e., prior to and on the same day of the next scheduled administration of CZP).
Biological: Certolizumab Pegol — Mothers who decided to continue on, or to start treatment with, Certolizumab Pegol (CZP) for an approved indication with their treating physician prior to participation into this study. The mother is responsible for procuring her own supply of commercial CZP. The CZP dose and administration schedule will be as per the locally approved label.
  Other Names: Cimzia®

SUMMARY:
The primary objectives of this study are to assess whether there is transfer of Certolizumab Pegol (CZP) into breast milk of lactating mothers who are receiving an established dosing regimen of CZP by evaluating the concentration of CZP in mature breast milk, and to calculate the daily infant dose of maternal CZP.

DETAILED DESCRIPTION:
The study will only include women who are receiving treatment with Certolizumab Pegol (CZP) for an approved indication in accordance with their treating physician, although this study is non-interventional regarding treatment with CZP, it is considered interventional due to the collection of breast milk from the lactating mothers.

ELIGIBILITY:
Inclusion Criteria:

* An IRB/IEC approved written Informed Consent form for participation of the maternal subject and her infant (for collection of infant demographic and AE data) is signed and dated by the subject. Where applicable, the written Informed Consent form with respect to the infant is also signed and dated by the holder of parental rights as designated by the maternal subject
* Subject is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the Investigator
* Subject is female and at least 18 years of age at the time of providing consent
* Subject has delivered term infant(s) (at least 37 weeks gestation)
* Subject is being treated with Certolizumab Pegol (CZP) per the current approved prescribing information
* The decision to treat with CZP or to breastfeed is made independently from and prior to the subject consenting to participate in this study
* Subject agrees to use only the emollient or nipple cream provided by the Sponsor for use during the Sampling Period as described per protocol
* Subject is at least 6 weeks postpartum
* Subject is on an established dosing regimen of CZP (at least the third dose of CZP since starting/restarting CZP)

Exclusion Criteria:

* Subject is pregnant or plans to become pregnant during the study
* Subject is taking a prohibited medication or has taken a prohibited medication Note: any subjects requiring antibiotics must be discussed with the Medical Monitor prior to enrollment
* Subject has history of chronic alcohol abuse or drug abuse in the last year
* In subjects who intend to breastfeed, the infant has any abnormality noted on physical examination that, in the opinion of the Investigator, may jeopardize or compromise the subject's ability to participate in this study
* Subject has any medical, obstetrical or psychiatric condition that, in the opinion of the Investigator, can jeopardize or would compromise the subject's ability to participate in this study or the outcome of the pregnancy (as applicable). Note: subjects with mastitis infection should not have samples collected until the infection is completely resolved
* Subject has history of breast implants, breast augmentation, or breast reduction surgery
* Subject has previously participated in this study
* Subject has participated in a study of an investigational medicinal product (IMP) (or a medical device) within the previous 30 days or 5 half-lives (whichever is longer) prior to Screening or is currently participating in another study of an IMP (or a medical device) unless the study is UCB UP0017 [NCT02019602] or a registry study
* Subject has received treatment with any biological therapeutic agent, or other anti-TNF agents with the exception of CZP, within 5 half-lives prior to obtaining the first sample
* Subject has a positive or indeterminate QuantiFERON®-TB GOLD In Tube test at Screening. In case of indeterminate result, a retest is allowed if time permits; 2 results of indeterminate require exclusion of the subject
* Subject with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent TB (LTB) infection. If tested within the 6 months prior to screening and test was negative for TB, and there is no change in the patient's clinical status, nor social, family, or travel history, there is no need for an additional TB testing at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- United States (3):
  - 7, Los Angeles, California
  - 1, Chapel Hill, North Carolina
  - 3, Durham, North Carolina
- Netherlands (2):
  - 500, Maastricht
  - 501, Rotterdam
- 20, Bern, Switzerland

REFERENCES:
- [Result] Clowse ME, Forger F, Hwang C, Thorp J, Dolhain RJ, van Tubergen A, Shaughnessy L, Simpson J, Teil M, Toublanc N, Wang M, Hale TW. Minimal to no transfer of certolizumab pegol into breast milk: results from CRADLE, a prospective, postmarketing, multicentre, pharmacokinetic study. Ann Rheum Dis. 2017 Nov;76(11):1890-1896. doi: 10.1136/annrheumdis-2017-211384. Epub 2017 Aug 16. PMID 28814432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2014 and concluded in December 2015.
Pre-assignment Details: The Participant Flow refers to the Safety Set which consisted of 18 mothers, who were screened and had received at least one dose of Certolizumab Pegol (CZP), but only 17 mothers entered the study (Enrollment number), as one subject was a screen failure.
Groups:
- Mothers (SS): This arm consisted of all participating mothers who had received at least 1 dose of Certolizumab Pegol (CZP).
Period: Screening Period
Arm/Group | Mothers (SS)
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1
Period: Sampling Period
Arm/Group | Mothers (SS)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all participating mothers who had received at least 1 dose of CZP.
Arm/Group | Mothers (SS)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  arithmetic mean (standard deviation) | 33.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 0
Description: Mature breast milk samples were collected predose on Day 0 of the Sampling Period (CZP dosing day) for all subjects.
Time Frame: Day 0
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all subjects with a valid CZP concentration measurement in breast milk with no important protocol deviations affecting the primary variable.
Measure: Median (Full Range); unit: µg/mL
Groups:
- Mothers CZP (PK-PPS) Q2W: This arm consisted of all mothers with a valid Certolizumab Pegol (CZP) concentration measurement in breast milk with no important protocol deviations affecting the primary variable, who were administered 200 mg CZP every 2 weeks (Q2W).
- Mothers CZP (PK-PPS) Q4W: This arm consisted of all mothers with a valid Certolizumab Pegol (CZP) concentration measurement in breast milk with no important protocol deviations affecting the primary variable, who were administered 400 mg CZP every 4 weeks (Q4W).
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | NA [NA to 0.0571] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

2. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 2
Description: Mature breast milk samples were collected on Day 2 of the Sampling Period for all subjects.
Time Frame: Day 2
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | NA [NA to 0.0686] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

3. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 4
Description: Mature breast milk samples were collected on Day 4 of the Sampling Period for all subjects.
Time Frame: Day 4
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | 0.03578 [NA to 0.0742] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

4. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 6
Description: Mature breast milk samples were collected on Day 6 of the Sampling Period for all subjects.
Time Frame: Day 6
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | 0.03739 [NA to 0.0758] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

5. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 8
Description: Mature breast milk samples were collected on Day 8 of the Sampling Period for all subjects.
Time Frame: Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | 0.03899 [NA to 0.0755] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

6. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 10
Description: Mature breast milk samples were collected on Day 10 of the Sampling Period for all subjects.
Time Frame: Day 10
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | NA [NA to 0.0685] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

7. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 12
Description: Mature breast milk samples were collected on Day 12 of the Sampling Period for all subjects.
Time Frame: Day 12
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | NA [NA to 0.0694] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

8. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 14
Description: Mature breast milk samples were collected (predose, as applicable for subjects receiving CZP 200 mg Q2W) on Day 14 of the Sampling Period for all subjects.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q2W | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 16 | 1
µg/mL | NA [NA to 0.0603] — NA = below limit of quantification. | NA [NA to NA] — NA = below limit of quantification.

9. Primary Outcome: The Concentration of Certolizumab Pegol (CZP) in Breast Milk on Day 28
Description: In subjects receiving CZP 400 mg Q4W, a mature breast milk sample were collected on or about Day 28, prior to the next scheduled administration of CZP.
Time Frame: Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Mothers CZP (PK-PPS) Q4W
Number analyzed (Participants) | 1
µg/mL | NA [NA to NA] — NA = below limit of quantification.

10. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 2
Description: Mature breast milk samples was collected on Day 2 of the Sampling Period for all subjects.
Time Frame: Day 2
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Groups:
- All Mothers (PK-PPS): This arm consisted of all mothers with a valid CZP concentration measurement in breast milk with no important protocol deviations affecting the primary variable.
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0 [0 to 0.0103]

11. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 4
Description: Mature breast milk samples was collected on Day 4 of the Sampling Period for all subjects.
Time Frame: Day 4
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0.005306 [0 to 0.0111]

12. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 6
Description: Mature breast milk samples was collected on Day 6 of the Sampling Period for all subjects.
Time Frame: Day 6
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0.005604 [0 to 0.0114]

13. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 8
Description: Mature breast milk samples was collected on Day 8 of the Sampling Period for all subjects.
Time Frame: Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0.005606 [0 to 0.0113]

14. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 10
Description: Mature breast milk samples was collected on Day 10 of the Sampling Period for all subjects.
Time Frame: Day 10
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0 [0 to 0.0103]

15. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 12
Description: Mature breast milk samples was collected on Day 12 of the Sampling Period for all subjects.
Time Frame: Day 12
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0 [0 to 0.0104]

16. Primary Outcome: The Calculated Daily Infant Dose of Certolizumab Pegol (CZP) in Breast on Day 14
Description: Mature breast milk samples was collected (pre-dose, as applicable for subjects receiving CZP 200 mg Q2W) on Day 14 of the Sampling Period for all subjects.
Time Frame: Day 14
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0 [0 to 0.00904]

17. Primary Outcome: The Calculated Infant Daily Dose of Certolizumab Pegol (CZP) in Breast Milk on Day 28
Description: In subjects receiving CZP 400 mg Q4W, a mature breast milk sample was collected on or about Day 28, prior to the next scheduled administration of CZP.
Time Frame: Day 28
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all subjects with a valid CZP concentration measurement in breast milk with no important protocol deviations affecting the primary variable. Measurement on day 28 applies to subjects on a CZP 400mg Q4W dosing regimen only.
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 1
mg/kg/day | 0 [0 to 0]

18. Primary Outcome: The Average Daily Infant Dose of Certolizumab Pegol (CZP) Over the Dosing Interval (14 or 28 Days)
Description: Mature breast milk samples will be collected (pre-dose, as applicable for subjects receiving CZP 200 mg Q2W) on Day 14 or on Day 28 of the Sampling Period for all subjects.
Time Frame: From Day 0 to Day 14 or 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | All Mothers (PK-PPS)
Number analyzed (Participants) | 17
mg/kg/day | 0.003503 [0 to 0.0104]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the whole study period (from Week 0 to Week 19)
Groups:
- SS-M: This arm consisted of all participating mothers who had received at least 1 dose of Certolizumab Pegol (CZP).
- SS-I: This arm consisted of all infants of mothers in the SS-M.
Arm/Group | SS-M | SS-I
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/17
Other Adverse Events (participants affected / at risk) | 9/18 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS-M (N=18) | SS-I (N=17)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS-M (N=18) | SS-I (N=17)
Exacerbation of Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Candida infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Galactostasis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4)
Lichen striatus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days